CLINICAL TRIAL: NCT05250206
Title: Evaluation of Ophthalmic Lenses for Myopia Management
Brief Title: Evaluation of the Efficacy in Decreasing Myopia Progression of the Proposed Ophthalmic Lens Prototypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indizen Optical Technologies, S.L.U. (Industry)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IOT-MIO-2018-01
Record Dates: First submitted 2022-02-03; First posted 2022-02-22 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axial lenght increase (Experimental): Children aged 5 to 12 with myopia up to -0.50 D, astigmatism and anisometropia under 1.50 D, and corrected visual acuity over 20/20 will be randomized to either the control group or treatment group. The myopia progression was evaluated by measuring axial length (AL) growth (IOL Master; Zeiss) over a period of one year.
  Interventions: Other: Myopia control lens

INTERVENTIONS:
Other: Myopia control lens — Evaluation of the efficacy in decreasing myopia progression of the proposed ophthalmic lens prototypes.

SUMMARY:
Evaluation of the efficacy in decreasing myopia progression of the proposed ophthalmic lens prototypes.

DETAILED DESCRIPTION:
A prospective, double-blind, randomized clinical trial (RCT) to analyze the effect of a new ophthalmic lens prototype on myopia progression. The follow-up period to evaluate the efficacy of the lens will be 3 years including a total of 5 visits.

The sample will consist of a group of 92 myopic children who will be randomly assigned to one of the treatment groups:

* Control group who will receive standard monofocal lenses.
* Treatment group who will wear a prototype lens based on peripheral positive defocus.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 to 12 years old
* Myopia (spherical equivalent with cycloplegic) ≤ -0.50D
* Astigmatism < 1.50D
* Anisometropia < 1.50D
* Best-corrected visual acuity ≥ 20/20

Exclusion Criteria:

* Patients who have received any previous treatment for myopia control, including the use of RPG contact lenses.
* Participants with ocular pathology such as retinal detachment.
* Participants using drugs that may affect pupillary size and accommodation or that produce effects on the ocular surface.
* Participants with systemic diseases that may affect vision.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasebe S, Jun J, Varnas SR. Myopia control with positively aspherized progressive addition lenses: a 2-year, multicenter, randomized, controlled trial. Invest Ophthalmol Vis Sci. 2014 Sep 30;55(11):7177-88. doi: 10.1167/iovs.12-11462. PMID 25270192
- [Background] Kanda H, Oshika T, Hiraoka T, Hasebe S, Ohno-Matsui K, Ishiko S, Hieda O, Torii H, Varnas SR, Fujikado T. Effect of spectacle lenses designed to reduce relative peripheral hyperopia on myopia progression in Japanese children: a 2-year multicenter randomized controlled trial. Jpn J Ophthalmol. 2018 Sep;62(5):537-543. doi: 10.1007/s10384-018-0616-3. Epub 2018 Aug 6. PMID 30083910
- [Background] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Lens: Standard spherocylindrical lenses.
- Treatment Lens: Lenses with a central zone that provides the patient's optimal prescription surrounded by a zone of positive defocus that increases progressively from the center to the periphery of the lens, in an asymmetrical manner between the different zones of the lens.
Period: Overall Study
Arm/Group | Control Lens | Treatment Lens
Started | 46 | 46
Completed | 34 | 35
Not Completed | 12 | 11

BASELINE CHARACTERISTICS:
Population: 92 children were enrolled and 23 of the participants did not complete the study. Thus, the final sample was 69 children.
Groups:
- Control Group: The control group consisted of 34 children using standard spherocylindrical lenses.
- Treatment Group: The treatment group included 35 children wearing a prototype lens with a central zone that provides the patient's optimal prescription surrounded by a zone of positive defocus that increases progressively from the center to the periphery of the lens, in an asymmetrical manner between the different zones of the lens.
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] — The age of the children who participated in the study ranged from 6.4 to 13.7 years
  years | 9.6 (1.8) | 10.4 (1.8) | 10.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 40
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Spanish children | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Axial Lenght Increase
Description: Axial length was measured with the IOL Master® optical biometer (Carl Zeiss Meditec, Jena, Germany) and axial length growth was calculated by subtracting the axial length measurement after one year of treatment and the axial length at the initial visit.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Myopia Control Lens: The control group consisted of 42 children using standard spherocylindrical lenses.
- Treatment Group: The treatment group included 41 children wearing a prototype lens with a central zone that provides the patient's optimal prescription surrounded by a zone of positive defocus that increases progressively from the center to the periphery of the lens, in an asymmetrical manner between the different zones of the lens.
Arm/Group | Myopia Control Lens | Treatment Group
Number analyzed (Participants) | 34 | 35
mm | 0.27 (0.23) | 0.37 (0.24)

ADVERSE EVENTS:
Time Frame: From baseline through 24 months of follow-up
Description: Adverse events were monitored continuously from baseline to study completion (24 months). Only participants who completed the study were included in the final safety analysis (n=69).
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT05250206/Prot_SAP_000.pdf